CLINICAL TRIAL: NCT01488695
Title: Comparison of GlideScope Groove to Macintosh Blade for Orotracheal Intubation With Double-Lumen Endotracheal Tube: a Randomised Controlled Trial
Brief Title: GlideScope Groove Versus Macintosh Blade for Double-Lumen Endotracheal Tube Intubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device withdrawn from the market
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Timothy Turkstra, Staff anesthesiologist and Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 18478
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Intubation, Intratracheal
Keywords: intubation; double lumen tube

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideScope Groove (Experimental): Patient will be intubated using the GlideScope Groove device.
  Interventions: Device: GlideScope Groove
- Control (Active Comparator): Control Group: Macintosh Blade
  Interventions: Device: Control: Macintosh blade

INTERVENTIONS:
Device: GlideScope Groove — GlideScope Groove
  Other Names: Verathon
  Arms: GlideScope Groove
Device: Control: Macintosh blade — Control: Patients will be intubated using the Macintosh blade
  Other Names: Mac 3, 4
  Arms: Control

SUMMARY:
A new GlideScope videolaryngoscope has been developed, which utilizes a track on the superior surface of the blade to guide the endotracheal tube, which is advanced in the track as opposed to "free-hand" along the inferior surface, where the camera is located. This new GlideScope can be used for double-lumen endotracheal tubes (DLT). The investigators hypothesize that this GlideScope will be easier to use than the Macintosh blade.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient booked for elective surgery requiring orotracheal intubation with a double lumen endotracheal tube.

Exclusion Criteria:

1. Any patient with cervical spine abnormalities.
2. Any patients with known or probable difficult airways.
3. Any patient requiring rapid sequence induction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Duration of Intubation | Day 1
  The intubation will be timed using a stopwatch.

SECONDARY OUTCOMES:
Number of intubation attempts | Day 1
  Number of intubation attempts
Number of failures to intubate | Day 1
  Number of failures to intubate
Use of external laryngeal pressure | Day 1
  Whether or not external laryngeal pressure was needed to facilitate tracheal intubation
Laryngoscopic grade distribution | Day 1
  Cormack and Lehane Grade observed during laryngoscopy
Presence of Sore throat | Day 3
  Sore throat will be graded on POD #2 as none, mild, moderate, or severe

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, Principal Investigator — University of Western Ontario, Canada
Locations (2):
- Canada (2):
  - London Health Sciences Center University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario